CLINICAL TRIAL: NCT05954819
Title: Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing, Department of Medical Nursing
Brief Title: Effect of Patient Education on Healthy Lifestyle Behaviors and Diabetes Self-management in Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Arzu Erkoc, Istanbul University - Cerrahpasa, Florence Nightingale Faculty of Nursing, Department of Medical Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC 2022/476
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2; Myocardial Infarction
Keywords: Diabetes; Patient education; Diabetes self-management; Myocardial infarction; Healthy lifestyle behaviors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planned patient education (Experimental): Pre-test data will be obtained by using the "Healthy Lifestyle Behaviors Scale" and "Diabetes Self-Management Scale". The participants will be individual education on myocardial infarction and diabetes by researcher. One month later, the posttest data will be obtained using "Healthy Lifestyle Behaviors Scale" and "Diabetes Self-Management Scale".
  Interventions: Other: Planned patient education
- Routine patient education (No Intervention): Pre-test data will be obtained by using "Healthy Lifestyle Behaviors Scale" and "Diabetes Self-Management Scale". No attempt will be made to participants by the researcher. Participants will undergo discharge training routinely administered by bedside nurses at the hospital. One month later, the posttest data will be obtained using "Healthy Lifestyle Behaviors Scale" and "Diabetes Self-Management Scale".

INTERVENTIONS:
Other: Planned patient education — Patients in the experimental group will be given about 30 minutes of patient education. After the training, a Patient Education Booklet containing Myocardial Infarction and Diabetes Education will be presented to the patients. Control group patients will not be given any training other than the hospital routine.
  Arms: Planned patient education

SUMMARY:
The purpose of this study is to determine the effect of planned education given to individuals with diabetes mellitus who had myocardial infarction on healthy lifestyle behaviors and diabetes self-management.

DETAILED DESCRIPTION:
Many coronary heart patients have diabetes. For this reason, it is thought that patients need education in order to gain healthy lifestyle behaviors and to provide self-management of diabetes, which is a major risk factor for coronary artery disease. When the literature was examined, no study could be found that focused on diabetes patients with myocardial infarction and emphasized the importance of patient education. It is thought that this study will make an important contribution in terms of patient education to be given to individuals with diabetes mellitus who have had myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* No advanced hearing and vision problems,
* Able to speak and understand Turkish,
* Easy to communicate,
* Literate,
* Agreeing to participate in the research voluntarily,
* Hospitalized due to myocardial infarction in the last month,
* Have stayed in the intensive care unit for at least 24 hours,
* No chest pain
* Patients who have been diagnosed with Type 2 Diabetes Mellitus for at least one year

Exclusion Criteria:

* Sedative or narcotic analgesic drug treatment,
* Use of antipsychotic medication
* Patients receiving Continous Positive Airway Pressure treatment,
* Patients with cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change of Healthy Lifestyle Behaviors | Change from Baseline Healthy Lifestyle Behaviors at 4 Weeks
  The Healthy Lifestyle Behaviors Scale, which consists of 52 items, has a total of 6 sub-dimensions: spiritual development, health responsibility, physical activity, nutrition, spiritual development, interpersonal relations and stress management.The overall score of the scale gives the healthy lifestyle behaviors score.
Change of Diabetes Self-Management | Change from Baseline Diabetes Self-Management at 4 Weeks
  The Diabetes Self-Management Scale, which consists of 19 questions in the scale that evaluate self-management in patients with type 2 diabetes. High scores on the scale indicate good self-management, and low scores indicate poor self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Erkoc, Study Director — Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing
Locations (1):
- Istanbul University-Cerrahpasa Florence Nightingale Faculty of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study is planned as a master's thesis. Data can be shared after the thesis is completed.
Time Frame: The data will become available after two years.
Access Criteria: Criteria is to refer to this study.